CLINICAL TRIAL: NCT02140645
Title: Association of Clinical Covariates With Non-insulin Diabetes Medication Initiation Using Electronic Medical Records (EMR)
Brief Title: Ascertainment of EMR-based Clinical Covariates Among Patients Receiving Oral and Non-insulin Injected Hypoglycemic Therapy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.162
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (6):
- Linagliptin1: T2DM patients initiating Linagliptin (DPP-4 comparison)
  Interventions: Drug: linagliptin
- Other DPP4: T2DM patients initiating a non-linagliptin DPP-4 inhibitor
- Linagliptin2: T2DM patients initiating Linagliptin (glitizaone comparison)
- Glitazones: T2DM patients initiating Thiazolidinediones (glitazones)
- Sulfonylurea: T2DM patients initiating any medication in the Sulfonylurea class
- Linagliptin3: T2DM patients initiating Linagliptin (Sulfonylurea comparison)

INTERVENTIONS:
Drug: linagliptin — non-randomized
  Groups: Linagliptin1

SUMMARY:
The objective of this study is to identify EMR-based clinical covariates and quantify their association with the prescribing of each specific type 2 diabetes (T2DM) medication under investigation. This will include an assessment of how well these covariates are captured through claims data proxies, and their potential to confound comparative research of T2DM medications.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Dispensing of an oral or non-insulin injected hypoglycemic medication between May 2011 and June 2012
* Diagnosis of type 2 diabetes mellitus
* Presence of electronic medical records (for the EMR-based subset)

Exclusion criteria:

* Age <18 at T2DM medication initiation
* Missing or ambiguous age or sex information
* At least one diagnosis of type 1 diabetes mellitus
* Less than 6 months enrolment in the database preceding the date of the first dispensing
* Prior use of the index drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients aged 18 or older, initiating antidiabetic treatment after at least 6 months of continuous enrollment
Sampling Method: Non-Probability Sample
Enrollment: 166613 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Existing data cohort design using data from the MarketScan database from May 2011 through December 2012. 492963 potential patients were identified in the database, but after removing patients who violated inclusion and exclusion criteria 166613 patients were actually analysed in the study.
Groups:
- Linagliptin 1: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication Linagliptin subjects matched to any other DPP-4 (Dipeptidyl peptidase-4 inhibitors).
- Any Other DPP-4: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication DPP-4 (Dipeptidyl peptidase-4 inhibitors).
- Linagliptin 2: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication Linagliptin subjects matched to pioglitazone.
- Pioglitazone: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication pioglitazone.
- Linagliptin 3: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication Linagliptin subjects matched to second generation sulfonylurea.
- Second Generation Sulfonylurea: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication second generation sulfonylurea.
Period: Overall Study
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Started | 5732 | 64695 | 4441 | 14363 | 3436 | 73946
Completed | 243 | 3041 | 205 | 530 | 150 | 3050
Not Completed | 5489 | 61654 | 4236 | 13833 | 3286 | 70896
Not completed — Not linked | 5489 | 61654 | 4236 | 13833 | 3286 | 70896

BASELINE CHARACTERISTICS:
Population: All patients who did not violate any inclusion/exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea | Total
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050 | 7219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (11.6) | 54.8 (11.2) | 55.2 (11.7) | 54.7 (11.1) | 54.7 (11.8) | 54.8 (11.7) | 54.9 (11.5)
Gender [Count of Participants; unit: Participants]
  Female | 118 | 1310 | 101 | 194 | 74 | 1332 | 3129
  Male | 125 | 1731 | 104 | 336 | 76 | 1718 | 4090

OUTCOME MEASURES:

1. Primary Outcome: Missing EMR (Electronic Medical Record) Characteristic: Smoking
Description: The missing EMR characteristic smoking defined as current, unknown, versus past/never smoker.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic smoking was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: All subjects in MarketScan cohort meeting inclusion/exclusion criteria. EMR-linked subset: From the study group we identified patients who have EMR data available.
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants
  Current | 9.1 | 7.6 | 10.7 | 7.9 | 11.3 | 9.4
  Past | 12.3 | 12.2 | 12.2 | 10.2 | 10.7 | 10.9
  Never | 32.9 | 35.5 | 32.7 | 30.8 | 34.7 | 33.3
  Unknown | 5.8 | 4.9 | 6.3 | 5.1 | 6.0 | 6.5
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.624 — The C-statistics can be between 0.5 and 1 and a value of 0.5 indicates that the model is no better than chance at making a prediction and a value of 1.0 indicates that the model perfectly identifies those within a group and those not

2. Primary Outcome: Missing EMR Characteristic: Duration of Diabetes
Description: The missing EMR characteristic duration of diabetes defined as >7, 5-6, 3-5, 1-3, <1 (in years) in duration.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic duration of diabetes was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants
  Less than 1 year | 11.9 | 13.7 | 12.7 | 11.1 | 16.0 | 15.4
  1.00-2.99 years | 11.5 | 14.2 | 11.2 | 10.0 | 12.7 | 13.6
  3.00-4.99 years | 7.8 | 7.8 | 7.8 | 8.3 | 7.3 | 8.4
  5.00-6.99 years | 4.9 | 5.1 | 3.9 | 5.7 | 4.0 | 4.8
  7+ years | 5.3 | 5.3 | 5.4 | 5.8 | 5.3 | 4.8
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistcs = 0.597 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Missing EMR Characteristic: Duration of Diabetes (Continuous)
Description: The missing EMR characteristic duration of diabetes defined as starting year/starting age of diabetes.
  Linear regression models were ran using a prioritized list of claims-based covariates as predictors and the value of select EMR-based clinical characteristics duration of diabetes as continuous outcomes.
  The estimated value represented is actually prediction accuracy defined by R-squared.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Months | 3.5 (3.7) | 3.1 (3.3) | 3.4 (3.7) | 3.5 (3.1) | 3.0 (3.4) | 2.9 (3.0)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; R-squared = 0.0858 — The R-squared can be between 0 and 1 and a value of 0 indicates that the model is no better than chance at making a prediction and a value of 1.0 indicates that the model perfectly identifies those within a group and those not

4. Primary Outcome: Missing EMR Characteristic: BMI (Body Mass Index)
Description: The missing EMR characteristic BMI defined as not obese, overweight, obese, severe obesity.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic BMI was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants
  Underweight | 0.4 | 0.1 | 0.5 | 0.0 | 0.7 | 0.1
  Normal | 2.1 | 3.9 | 2.0 | 3.4 | 2.7 | 4.0
  Overweight | 11.5 | 11.8 | 13.7 | 15.5 | 10.7 | 14.0
  Obese | 35.4 | 35.1 | 35.1 | 29.6 | 36.0 | 34.2
  Severe Obesity | 16.5 | 15.5 | 16.1 | 10.9 | 16.0 | 15.4
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.623 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Missing EMR Characteristic: BMI (Continuous)
Description: The missing EMR characteristic BMI is BMI value. Linear regression models were ran using a prioritized list of claims-based covariates as predictors and the value of select EMR-based clinical characteristics BMI as continuous outcomes.
  The estimated value represented is actually prediction accuracy defined by R-squared.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Kg/m^2 | 36.3 (8.5) | 35.5 (8.0) | 36.1 (8.8) | 34.2 (7.0) | 36.6 (9.2) | 35.1 (7.8)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; R-squared = 0.1753 — [estimate comment as in outcome 3, analysis 1]

6. Primary Outcome: Missing EMR Characteristic: HbA1c (Hemoglobin A1c (Glycosylated Hemoglobin))
Description: The missing EMR characteristic HbA1c defined as value in 6 months prior to and including index date.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic HbA1c was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage | 8.2 (1.4) | 8.6 (1.9) | 8.3 (1.4) | 9.0 (2.2) | 8.0 (1.5) | 8.8 (2.0)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.699 — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Missing EMR Characteristic: eGFR (Glomerular Filtration Rate)
Description: The missing EMR characteristic eGFR defined as value in 6 months prior to and including index date.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic eGFR was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Upto 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/min per 1.73 m^2
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
ml/min per 1.73 m^2 | 103.8 (19.2) | 107.0 (18.0) | 104.9 (18.7) | 108.7 (19.3) | 105.5 (18.5) | 106.8 (18.7)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.683 — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Missing EMR Characteristic: Total Cholesterol
Description: The missing EMR characteristic total cholesterol defined as value in 6 months prior to and including index date.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic total cholesterol was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
mg/dl | 188.8 (59.7) | 177.6 (47.0) | 189.7 (62.9) | 185.8 (58.8) | 194.6 (53.1) | 185.8 (50.8)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.757 — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Missing EMR Characteristic: Systolic BP (Blood Pressure)
Description: The missing EMR characteristic systolic BP defined as value in 6 months prior to and including index date.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic systolic BP was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
mmHg | 130.2 (16.3) | 129.7 (15.7) | 131.0 (16.1) | 131.5 (17.2) | 131.2 (17.3) | 131.3 (17.0)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.618 — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Missing EMR Characteristic: Diastolic BP
Description: The missing EMR characteristic diastolic BP defined as value in 6 months prior to and including index date.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic diastolic BP was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
mmHg | 79.5 (10.6) | 78.8 (10.0) | 80.0 (10.2) | 79.3 (10.6) | 80.0 (10.5) | 79.6 (10.5)
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.618 — [estimate comment as in outcome 1, analysis 1]

11. Primary Outcome: Binary EMR Characteristic: Neuropathy
Description: The missing EMR characteristic neuropathy defined as participants with any note of diabetic neuropathy.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic neuropathy was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants | 9.9 | 10.0 | 10.7 | 11.3 | 12.0 | 11.0
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.733 — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Binary EMR Characteristic: Nephropathy
Description: The missing EMR characteristic nephropathy defined as participants with any note of diabetic nephropathy.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic nephropathy was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Upto 20 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants | 5.8 | 3.2 | 5.9 | 4.3 | 4.7 | 3.0
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.827 — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Binary EMR Characteristic: Retinopathy
Description: The missing EMR characteristic retinopathy defined as participants with any note of diabetic retinopathy.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic retinopathy was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants | 1.2 | 1.9 | 1.0 | 2.8 | 1.3 | 1.7
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.801 — [estimate comment as in outcome 1, analysis 1]

14. Primary Outcome: Binary EMR Characteristic: Pancreatitis
Description: The missing EMR characteristic pancreatitis defined as participants with any note of prior pancreatitis.
  The associations between claims-based covariates and missingness on EMR characteristics were investigated by estimating a logistic regression model (and multinomial logistic regression, depending on the number of categories for the EMR characteristic) for each EMR characteristic where an indicator for missing the EMR characteristic pancreatitis was the dependent variable and all claims-based covariates were included as independent variables.
  The estimated value represented is actually prediction accuracy defined by C-statistics.
Time Frame: Up to 20 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linagliptin 1 | Any Other DPP-4 | Linagliptin 2 | Pioglitazone | Linagliptin 3 | Second Generation Sulfonylurea
Number analyzed (Participants) | 243 | 3041 | 205 | 530 | 150 | 3050
Percentage of participants | 0.8 | 0.5 | 1.0 | 0.2 | 0.7 | 0.5
Statistical Analysis 1: Comparison: Linagliptin 1 vs Any Other DPP-4 vs Linagliptin 2 vs Pioglitazone vs Linagliptin 3 vs Second Generation Sulfonylurea; Test type: Superiority or Other; C-statistics = 0.836 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Serious and other (non-serious) adverse events were not of interest in this study and therefore were not collected or assessed as part of the study, in addition individual patient data is not available therefore adverse event data is not presented.
Groups:
- MarketScan: Patients had a recorded diagnosis of type 2 diabetes mellitus (T2DM) using an oral and non-insulin injected glucose-lowering medication identified from the MarketScan database.
Arm/Group | MarketScan
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.